CLINICAL TRIAL: NCT03416725
Title: Evaluation of Prognostic Factors and Middle Ear Risk Index in Tympanoplasty
Brief Title: Evaluation of Prognostic Factors in Tympanoplasty
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, asmaa.nabil, Principal investigator, Assiut University
Other Study IDs: MERI
Record Dates: First submitted 2018-01-12; First posted 2018-01-31 (Actual); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Tympanic Membrane Perforation
MeSH Terms: conditions — Tympanic Membrane Perforation | interventions — Otoscopes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with chronic suppurative otitis media.: patients of the age group 18-60 years with Chronic suppurative otitis media (CSOM) planned for tympanoplasty.
  Interventions: Device: Otoscope

INTERVENTIONS:
Device: Otoscope — Otoscopic examination will be done to find the presence or absence of perforation, granulation tissue and cholesteatoma.

SUMMARY:
Tympanoplasty is the surgical operation performed for the reconstruction of the eardrum and/or the ossicles. Tympanoplasty is classified into five different types, originally described by Horst Ludwig Wullstein. 1,2 Type 1 involves repair of the tympanic membrane alone, when the middle ear is normal. A type 1 tympanoplasty is synonymous to myringoplasty, Type 2 involves repair of the tympanic membrane and middle ear in spite of slight defects in the middle ear ossicles, Type 3 when mallus and incus are absent graft place directly on stapes head., Type 4 describes a repair when the stapes foot plate is movable, but the crura are missing. The resulting middle ear will only consist of the Eustachian tube and hypotympanum, Type 5 is a repair involving a fixed stapes footplate.

There are various prognostic factors reported in the literature that may influence the surgical success of tympanoplasty.

DETAILED DESCRIPTION:
Some studies report significance for some of these factors whereas others report the contrary. The reported incidence of surgical success of tympanoplasty ranges from 60% to 99% in adults Belluci described four separate stages for prognosis of tympanoplasty 4 according to otorrhea

. Austin proposed a prognostic stratification according to disease categories, stage categories, and disease descriptors.

Black introduced the surgical, prosthetic, infection, tissues, and eustachian tube system (SPITE), and more recently Kartush developed middle ear risk index (MERI).

Smoking is added as a middle ear risk. Furthermore, cholesteatoma and granulation tissue or effusion risk value has been increased in MERI 2001.

Prognostic factors such as age, sex, presence of systemic diseases, location and size of perforation, duration of dry period, presence of myringosclerosis, presence of septal and conchal pathology, operation type, and status of the opposite ear and middle ear risk index were investigated. 9

ELIGIBILITY:
Inclusion Criteria:

* patients of the age group 18-60 years with Chronic suppurative otitis media (CSOM) planned for tympanoplasty.

Exclusion Criteria:

* Patients with otomycosis, septic foci such as sinusitis which can influence the outcome of tympanoplasty were excluded from the study

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: People with CSOM planning to make tympanoplasty
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2018-03-01 (Estimated); Primary Completion 2019-03-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of prognostic factors in tympanoplasty to predict the outcome of the surgical management whenever done. | One year
  Prognostic factors such as age, sex, presence of systemic diseases, location and size of perforation, duration of dry period, presence of myringosclerosis, presence of septal and conchal pathology and status of the opposite ear and middle ear risk index will be investigated.
Evaluation of middle ear risk index in tympanoplasty | One year
  Each risk parameter will take a numerical value; Ear discharge: 0-3, Perforation: 0-2, Cholesteotoma: 0-2, Ossicular chain status: 0-4, Middle ear granulation and history of previous surgery: 0-2. Now newly, smoking is also included as a risk parameter. The MERI will be evaluated. The patients will be categorized into those with mild (0-3), moderate(4-6) and severe(≥7) MERI

REFERENCES:
- [Background] Kartush JM. Ossicular chain reconstruction. Capitulum to malleus. Otolaryngol Clin North Am. 1994 Aug;27(4):689-715. PMID 7984370
- [Background] Becvarovski Z, Kartush JM. Smoking and tympanoplasty: implications for prognosis and the Middle Ear Risk Index (MERI). Laryngoscope. 2001 Oct;111(10):1806-11. doi: 10.1097/00005537-200110000-00026. PMID 11801949
- [Background] WULLSTEIN H. Theory and practice of tympanoplasty. Laryngoscope. 1956 Aug;66(8):1076-93. doi: 10.1288/00005537-195608000-00008. No abstract available. PMID 13358259